CLINICAL TRIAL: NCT02806518
Title: Evaluation of Dynamic Infrared Thermography as an Alternative to CT Angiography for Perforator Mapping in Breast Reconstruction
Brief Title: Dynamic Infrared Thermography as an Alternative to CT Angiography
Acronym: DIRT
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Other Study IDs: 2009/17(REK)
Record Dates: First submitted 2016-06-15; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: DIEP; Computed Tomography; Doppler; Thermography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women scheduled for DIEP: Women scheduled for DIEP breast reconstruction after mastectomy due to breast cancer are examined with DIRT, hand-held Doppler and CTA
  Interventions: Procedure: DIRT

INTERVENTIONS:
Procedure: DIRT — An infrared camera is used to capture video sequences of thermal images before, during and after exposure of the lower abdomen to a cold challenge.

SUMMARY:
Dynamic infrared thermography (DIRT) is an imaging method that does not require ionizing radiation or contrast injection. The study evaluates if DIRT can be an alternative to computed tomographic angiography (CTA) in perforator mapping. DIRT findings are compared with hand-held Doppler, CTA and intraoperative findings.

DETAILED DESCRIPTION:
In deep inferior epigastric perforator flap (DIEP) breast reconstruction the blood supply to the DIEP flap is reestablished by anastomosing the perforator to the internal mammary vessels. The selected perforator is crucial for flap survival as it is the only source of blood supply to the flap. CTA allows for precise anatomical description of the origin of perforators, their intramuscular course and point of fascia penetration but expose the patient to ionizing radiation and an intravenous contrast medium.

DIRT is an imaging method that does not require ionizing radiation or contrast injection. The study evaluates if DIRT can be an alternative to CTA in perforator mapping. The study is performed in a hospital where DIRT and CTA have been established preoperative imaging methods that have been used for several years as routine examinations for all DIEP breast reconstruction patients.

25 patients scheduled for secondary breast reconstruction with a DIEP flap are included. Preoperatively, the lower abdomen is examined with hand-held Doppler, DIRT and CTA. Arterial Doppler sound locations are marked on the skin.

DIRT examination involves rewarming of the abdominal skin after a mild cold challenge. The locations of hot spots on DIRT are compared with the arterial Doppler sound locations. The rate and pattern of rewarming of the hot spots are analyzed. Multiplanar CT reconstructions are used to see if hot spots are related to perforators on CTA and intraoperative findings.

When intraoperative findings confirm that a useful perforator is located at the same localization as indicated with DIRT, this perforator is used for DIEP breast reconstruction. Postoperatively the surgical outcome and possible complications related to the selected perforator are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for breast reconstruction with DIEP flap

Exclusion Criteria:

* Prior breast reconstruction / abdominal flap surgery

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women scheduled for DIEP breast reconstruction after mastectomy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Comparison of DIRT with hand-held Doppler, CTA and intraoperative findings | Preoperative
  Comparison of localization of hot spots on DIRT and arterial Doppler sound locations, perforators on CTA and useful perforators seen intraoperatively

SECONDARY OUTCOMES:
Surgical results | First postoperative month
  Registration of flap failure (patients operated with DIEP based on perforator indicated with DIRT)

CONTACTS AND LOCATIONS:
Overall Officials: Sven Weum, MD PhD, Principal Investigator — Associate Professor
Locations (1):
- University Hospital of North Norway, Tromsø, Trom, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cina A, Salgarello M, Barone-Adesi L, Rinaldi P, Bonomo L. Planning breast reconstruction with deep inferior epigastric artery perforating vessels: multidetector CT angiography versus color Doppler US. Radiology. 2010 Jun;255(3):979-87. doi: 10.1148/radiol.10091166. Epub 2010 Apr 14. PMID 20392982
- [Background] Mathes DW, Neligan PC. Current techniques in preoperative imaging for abdomen-based perforator flap microsurgical breast reconstruction. J Reconstr Microsurg. 2010 Jan;26(1):3-10. doi: 10.1055/s-0029-1244806. Epub 2009 Dec 18. PMID 20024888
- [Background] Blondeel PN, Beyens G, Verhaeghe R, Van Landuyt K, Tonnard P, Monstrey SJ, Matton G. Doppler flowmetry in the planning of perforator flaps. Br J Plast Surg. 1998 Apr;51(3):202-9. doi: 10.1016/s0007-1226(98)80010-6. PMID 9664879
- [Background] de Weerd L, Mercer JB, Weum S. Dynamic infrared thermography. Clin Plast Surg. 2011 Apr;38(2):277-92. doi: 10.1016/j.cps.2011.03.013. PMID 21620152
- [Background] de Weerd L, Weum S, Mercer JB. The value of dynamic infrared thermography (DIRT) in perforatorselection and planning of free DIEP flaps. Ann Plast Surg. 2009 Sep;63(3):274-9. doi: 10.1097/SAP.0b013e3181b597d8. PMID 19700958
- [Derived] Weum S, Mercer JB, de Weerd L. Evaluation of dynamic infrared thermography as an alternative to CT angiography for perforator mapping in breast reconstruction: a clinical study. BMC Med Imaging. 2016 Jul 15;16(1):43. doi: 10.1186/s12880-016-0144-x. PMID 27421763